CLINICAL TRIAL: NCT03591900
Title: Evaluation of Continuous Blood Glucose Monitoring Method for Detection of Alterations in Glucose Homeostasis in Beta Thalassemia Patients
Brief Title: The Use of CGMS to Detect Alterations of Blood Glucose in Thalassemic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Amira Abd el moneam, Professor of pediatrics, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: Pediatric hospital ASU
Record Dates: First submitted 2016-06-21; First posted 2018-07-19 (Actual); Last update posted 2018-07-19 (Actual); Status verified 2018-07

CONDITIONS: Diabetes; Prediabetes; B-Thalassemia
Keywords: early diabetes; prediabetes; continuous glucose monitoring system; detection
MeSH Terms: conditions — Diabetes Mellitus; Prediabetic State; beta-Thalassemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- daibetic thalassemic patients on SC insulin (Active Comparator): A pilot study will be done on 20 patients with abnormal glucose tolerance which will include:
  A-Continuous glucose monitoring system (CGMS) : A glucometer will be given to each patient and will be asked to measure blood glucose before meals and snacks and record the valus in the CGMS for better calibration (Khammar A et al., 2009).
  B-Therapeutic intervention:
  Thalassemia patients who proved to have diabetes according to the ADA criteria will be put on sc insulin
  Interventions: Device: insulin pump/CGMS
- daibetic thalassemic patients on insulin pump (Active Comparator): A pilot study will be done on 20 patients with abnormal glucose tolerance which will include:
  A-Continuous glucose monitoring system (CGMS) : A glucometer will be given to each patient and will be asked to measure blood glucose before meals and snacks and record the valus in the CGMS for better calibration (Khammar A et
  B-Therapeutic intervention:
  Thalassemia patients who proved to have diabetes according to the ADA criteria will be put on insulin pump
  Interventions: Device: insulin pump/CGMS

INTERVENTIONS:
Device: insulin pump/CGMS — A-Continuous glucose monitoring system (CGMS) : A glucometer will be given to each patient and will be asked to measure blood glucose before meals and snacks and record the valus in the CGMS for better calibration (Khammar A et al., 2009).
  B-Therapeutic intervention:
  Thalassemia patients who proved to have diabetes according to the ADA criteria will be subjected to
  • Insulin pump will be tried in each diabetic thalassemic patient versus conventional insulin therapy(Bruttomesso D et al., 2009).

SUMMARY:
The aim of the study is to:

* Assess the pattern of glucose homeostasis in patients with B thalassemia .
* To detect early impairment in glucose metabolism and prediabetic state in B thalassemia patients using continuous glucose monitoring system.
* To study the prevalence and type of DM in B thalassemia patients.
* A comparative study of standard insulin therapy compared to insulin pump therapy in thalassemic diabetic patients will be done.

The study will include screening of 200 children and adolescents who are regularly attending the Hematology Oncology Clinic and fulfilling the inclusion criteria for abnormalities of glucose homeostasis.

A pilot study will be done on 15 patients with abnormal glucose tolerance which will include:

A-Continuous glucose monitoring system (CGMS) : A glucometer will be given to each patient and will be asked to measure blood glucose before meals and snacks and record the valus in the CGMS for better calibration .

B-Therapeutic intervention:

Thalassemia patients who proved to have diabetes according to the ADA criteria will be subjected to

• Insulin pump will be tried in each diabetic thalassemic patient versus conventional insulin therapy.

DETAILED DESCRIPTION:
β-thalassemia is a worldwide distributed monogenic red cell disorder, characterized by the absence or reduced β-globin chain synthesis (De Franceschi et al.,2013).

Approximately 7% of the global population is carrier of such disorders, and 300,000-400,000 babies with severe forms of these diseases are born each year (Weatherall, 2005; Modell et al., 2008). Severe hereditary hemoglobin disorders of red cells occur at highest frequency in tropical regions.

Hemoglobinopathies constitute the single most common monogenic defect worldwide, and among hemoglobin disorders, the thalassemias prominently contribute to (Weatherall et al., 2001; de Franceschi et al., 2011). β-thalassemias (β-thal) are characterized by the presence of mutations on beta-globin gene resulting in the absence or reduced synthesis of β-globin chains.

Glucose metabolism disturbances, among other endocrinopathies, are a common feature of β -thalassaemia . Pancreatic iron overload and diabetes mellitus (DM) are common in thalassemia major patients. However, the relationship between iron stores and glucose disturbances is not well defined (Leila et al., 2012).

The etiology of DM in β -thalassemia is suggested to be due to the effect of iron overload on the different tissues controlling the carbohydrate homeostatic mechanisms; including the pancreas and liver. However, controversy about the etiology of this glycemic abnormality still exists (Weinberg 2007).

Both insulin deficiency and insulin resistance are reported in patients with β -thalassemia. Suggested risk factors for development of DM in patients with β -thalassemia include old age, increased amount of blood transfusion, high serum ferritin level, family history of DM, hepatic impairment, and genetic modifiers of iron overload( Cario et al., 2003;Suvarna , et al., 2006; Weinberg 2007).

Patients with DM had significantly impaired insulin sensitivity and insulin release (Bergman et al., 2010). Traditionally, insulin deficiency and long-standing insulin resistance (De Sanctis et al, 1988; Pappas et al, 1996) that result from direct toxic damage by iron to pancreatic-beta cells are thought to be the main underlying mechanisms leading from mild glucose intolerance to overt diabetes. As these endocrine complications result from chronic iron overload, they are much more common in patients whose chelation therapy is insufficient ( Farmaki et al., 2006).

Greater chelation options have improved survival (Chouliaras et al., 2011); however many patients still carry dangerous extrahepatic iron burdens. As patients live longer, cumulative iron-mediated toxicity compounded by natural aging makes diabetes a significant clinical problem.

Pancreatic iron loading in thalassemia major patients begins in early childhood, and the overall prevalence of diabetes mellitus (DM) ranges from 6.4% to 14.1% on cross-sectional studies (Borgna-Pignatti et al., 2004; Vogiatzi et al., 2009). Both insulin resistance and decreased insulin secretion contribute to diabetes in thalassemia major patients. (Angelopoulos et al., 2006; Cario et al., 2003; Hafez, 2009).

Diabetes prevalence in thalassemia has been shown to correlate with serum ferritin (Jaruratanasirikul et al., 2008; Siklar et al., 2008 ), with hepatitis C infection (Chern , 2001; Sougleri et al., 2001;Mowla et al., 2004) and with pancreatic and cardiac iron (Au et al., 2007; Matter et al., 2010).

Insulin pump therapy in the form of continuous subcutaneous insulin infusion (CSII) was introduced in the 1970s and turned out to ensure better metabolic control of diabetes compared to traditional insulin therapy approaches. It is currently considered to be the optimal method of insulin administration, since it imitates the pancreatic activity in the best possible way, ensures precise dosage, and at the same time offers a high level of ease and comfort (Bruttomesso D et al., 2009; Danne T et al., 2008).

Compared to the traditional methods of insulin therapy by means of multiple daily insulin injections (MDI), CSII can significantly decrease glycated hemoglobin (HbA1C), reduce 24-hour glucose variability, decrease incidence of severe hypoglycemia, and eliminate dawn phenomenon. Moreover, the use of CSII is associated with improved quality of life and precise insulin administration with respect to physical effort and diet(Jeitler K et al., 2008; Phillip M et al., 2007).

A long-term effect of CSII on the control of diabetes mellitus in thalassemics needs to be explained (Hammond P, 2004).

Aim of the work

The aim of the study is to:

* Assess the pattern of glucose homeostasis in patients with B thalassemia .
* To detect early impairment in glucose metabolism and prediabetic state in B thalassemia patients using continuous glucose monitoring system.
* To study the prevalence and type of DM in B thalassemia patients.
* A comparative study of standard insulin therapy compared to insulin pump therapy in thalassemic diabetic patients will be done.

Patients and methods

Subjects:

The study will include screening of 200 children and adolescents who are regularly attending the Hematology Oncology Clinic and fulfilling the inclusion criteria for abnormalities of glucose homeostasis. ADA criteria for diagnosing diabetes mellitus & impaired glucose tolerance (American Diabetes Association, 2013)

1. Diabetes symptoms (ie polyuria, polydipsia and unexplained weight loss) plus

   * a random venous plasma glucose concentration ≥126 mg/dl (7.0 mmol/l) or
   * a fasting plasma glucose concentration ≥126 mg/dl (7.0 mmol/l) (whole blood > 6.1mmol/l) or
   * two hour plasma glucose concentration ≥200 mg/dl (11.1 mmol/l). two hours after 75g anhydrous glucose in an oral glucose tolerance test (OGTT).
2. With no symptoms diagnosis should not be based on a single glucose determination but requires confirmatory plasma venous determination. At least one additional glucose test result on another day with a value in the diabetic range is essential, either fasting, from a random sample or from the two hour post glucose load. If the fasting or random values are not diagnostic the two hour value should be used

   * Impaired Glucose Tolerance (IGT) is a stage of impaired glucose regulation (Fasting plasma glucose < 7.0 mmol/ and OGTT two hour value > 7.8mmol/l but < 11.1 mmol/l).
   * Impaired Fasting Glycaemia (IFG) has been introduced to classify individuals who have fasting glucose values above the normal range but below those diagnostic of diabetes. (Fasting plasma glucose > 6.1 mmol/l but < 7.0 mmol/l). American Diabetes Patients proved to be diabetics according to the ADA criteria will be subjected to therapeutic intervention.

An informed consent will be obtained from each patient or his legal guardian before enrollement in the study.

A- Screening and recruitment stage

All included patients will be subjected to the following:

1. Detailed medical history taking with special stress on:

   * Demographic data (name, age, sex, consanguinity and socioeconomic class).
   * Age of diagnosis of thalassemia and disease duration.
   * Transfusion history:

     * Age of first transfusion.
     * Amount of blood in each transfusion.
     * Type of transfused PRBCs (filtered, washed, untreated).
     * Frequency of transfusion.
     * Calculation of transfusion index (packed red cell per body weight in Kg per year).
   * Iron chelation therapy:Type, dose, duration, complications and compliance to chelation therapy. Compliance will be assessed by reviewing patient self-report of dose-taking and the appropriate number of doses taken during each day will be checked by prescription refills and pill count (Claxton et al., 2001).
   * History of spleenectomy.
   * History of viral hepatitis ( hepatitis B and C virus).
2. Thorough clinical examination laying stress on:

   * Assessment of anthropometric measures including weight in kilograms (Kg) and height in centimeters (cm) and plotting them on the age- and sex-standard percentiles according to Egyptian growth charts (Diabetic endocrine and metabolic pediatric unit, 2003). Body mass index (BMI) will be measured as kg/m2. (Guldiken et al., 2007).
   * Measurement of vital data including heart rate and blood pressure.
   * BMI: simple index of weight-for-height that is commonly used to classify underweight, overweight and obesity. It is calculated as the weight in kilograms divided by the square of the height in meters( Kg/m2). (WHO, 1995).
   * Complete examination including cardiac, chest, abdominal and neurological examination.
   * Assessment of sexual maturity using Tanner score (Vichinsky et al., 2008):

   Delayed puberty and hypogonadism: Defined as absence of sexual characteristics in girls above the age of 13 years and a testicular volume < 4ml in boys above the age of 14 years. Arrested puberty is the non-progression of puberty for a period of 12 months. (Arya et al., 2005)
3. Laboratory investigations including:

   * Complete blood picture (CBC): using Sysmex XT-1800i (Sysmex, Japan) with examination of Leishman-stained smears for red blood cells (RBC) morphology and differential white blood cell (WBC) count.
   * Peripheral blood staining: by brilliant cresyl blue and examination of a smear for reticulocytic count
   * Qualitative and quantitative hemoglobin analysis: at time of diagnosis collected from follow up sheets of patients.
   * Hb electrophoresis to ensure diagnosis of B thalassemia.
   * Measurement of serum ferritin(Soliman AT, et al.; 2013).
   * Measurement of fasting C peptide.
   * Measurement of random and fasting plasma glucose level(American Diabetes Association, 2013).
   * Oral glucose tolerance test (Thennadil SN et al., 2001).

A pilot study will be done on 15 patients with abnormal glucose tolerance which will include:

A-Continuous glucose monitoring system (CGMS) : A glucometer will be given to each patient and will be asked to measure blood glucose before meals and snacks and record the valus in the CGMS for better calibration (Khammar A et al., 2009).

B-Therapeutic intervention:

Thalassemia patients who proved to have diabetes according to the ADA criteria will be subjected to

• Insulin pump will be tried in each diabetic thalassemic patient versus conventional insulin therapy(Bruttomesso D et al., 2009).

ELIGIBILITY:
Inclusion Criteria:

1. Patients with B-thalassemia as confirmed by qualitative and quantitative analysis of hemoglobin using high performance liquid chromatography ( HPLC) & reticulocytic count ( Wethers, 2000; Fung et al., 2008).
2. Patients with B-thalassemia aged less than 20 years.
3. Patients with B-thalassemia on regular blood transfusion.
4. Patients with B-thalassemia iron chelation therapy.
5. Patients with s. ferritin >1000(Soliman AT, et al.; 2013

Exclusion Criteria:

1. Alpha thalassemia and sickle thalassemia patients.
2. Patients with other endocrine abnormalities.
3. Patients with family history of DM or other systemic illness.
4. Patients with other hereditary diseases.

Max Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Actual)
Dates: Start 2014-04; Primary Completion 2016-06 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
number of thalassemic patients with impaired glucose tolerance | 2 years
  to find out the number of patients with thalassemia major having impaired glucose tolerance

SECONDARY OUTCOMES:
number of thalassemic patients with diabetes mellitus | 2 years
  to find out the number of patients with thalassemia major having diabetes mellitus
control of diabetic thalassemic patients on insulin pump | 2 years
  to compare the use of conventional insulin therapy to insulin pump in diabetic thalassemic patients